CLINICAL TRIAL: NCT03392532
Title: Axis Orientation Comparison of Two Silicone Hydrogel Toric Contact Lenses
Brief Title: Comparison of Two Silicone Hydrogel Toric Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: CLC127-C001
Record Dates: First submitted 2018-01-02; First posted 2018-01-08 (Actual); Results first posted 2019-01-29 (Actual); Last update posted 2019-01-29 (Actual); Status verified 2019-01

CONDITIONS: Astigmatism
Keywords: Astigmatism; Axis orientation
MeSH Terms: conditions — Astigmatism

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- AOHG toric, then AO toric (Other): Lotrafilcon B toric contact lenses with HYDRAGLYDE, followed by lotrafilcon B toric contact lenses, as randomized. Each product worn in both eyes for approximately 30 minutes, with a 30-45 minute washout between the removal of Pair 1 and insertion of Pair 2.
  Interventions: Device: Lotrafilcon B toric contact lenses with HYDRAGLYDE; Device: Lotrafilcon B toric contact lenses
- AO toric, then AOHG toric (Other): Lotrafilcon B toric contact lenses, followed by lotrafilcon B toric contact lenses with HYDRAGLYDE, as randomized. Each product worn in both eyes for approximately 30 minutes, with a 30-45 minute washout between the removal of Pair 1 and insertion of Pair 2.
  Interventions: Device: Lotrafilcon B toric contact lenses with HYDRAGLYDE; Device: Lotrafilcon B toric contact lenses

INTERVENTIONS:
Device: Lotrafilcon B toric contact lenses with HYDRAGLYDE — Silicone hydrogel soft contact lenses for astigmatism
  Other Names: AIR OPTIX® plus HYDRAGLYDE® for Astigmatism contact lenses; AOHG for Astigmatism
Device: Lotrafilcon B toric contact lenses — Silicone hydrogel soft contact lenses for astigmatism
  Other Names: AIR OPTIX® for Astigmatism contact lenses; AO for Astigmatism

SUMMARY:
The purpose of this research study is to compare the performance of two different types of Alcon soft toric study contact lenses to obtain information on study lens orientation.

ELIGIBILITY:
Inclusion Criteria:

* Successful wear of soft contact lenses for vision correction in both eyes during the past 3 months for a minimum of 3 days per week and 8 hours per day
* Astigmatism
* Requires contact lenses
* Best corrected visual acuity of 20/25 or better in each eye
* Other protocol-specified inclusion criteria may apply

Exclusion Criteria:

* Any eye condition that contraindicates contact lens wear, as determined by the Investigator
* Any eye surgery that contraindicates contact lens wear, as determined by the Investigator
* Other protocol-specified exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2018-01-04 (Actual); Primary Completion 2018-01-26 (Actual); Study Completion 2018-01-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alcon, A Novartis Division, Study Director — Alcon, A Novartis Division
Locations (1):
- Alcon Investigative Site, Johns Creek, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from one investigative site located in the US.
Pre-assignment Details: This reporting group includes all enrolled subjects (36).
Groups:
- AOHG Toric, Then AO Toric: Lotrafilcon B toric contact lenses with HYDRAGLYDE®, followed by lotrafilcon B toric contact lenses, as randomized. Each product worn in both eyes for approximately 30 minutes, with a 30-45 minute washout between the removal of Pair 1 and insertion of Pair 2.
- AO Toric, Then AOHG Toric: Lotrafilcon B toric contact lenses, followed by lotrafilcon B toric contact lenses with HYDRAGLYDE®, as randomized. Each product worn in both eyes for approximately 30 minutes, with a 30-45 minute washout between the removal of Pair 1 and insertion of Pair 2.
Period: Period 1, FIrst 30 Minutes of Wear
Arm/Group | AOHG Toric, Then AO Toric | AO Toric, Then AOHG Toric
Started (As randomized) | 18 | 18
Completed | 18 | 18
Not Completed | 0 | 0
Period: Period 2, Second 30 Minutes of Wear
Arm/Group | AOHG Toric, Then AO Toric | AO Toric, Then AOHG Toric
Started (As randomized) | 18 | 18
Completed | 18 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: This analysis population includes all randomized subjects exposed to any study lenses evaluated in this study (Full Analysis Set).
Groups:
- Overall: Lotrafilcon B toric contact lenses with HYDRAGLYDE® and lotrafilcon B toric contact lenses worn during Period 1 and Period 2 in a crossover assignment
Arm/Group | Overall
Number analyzed (Participants) | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.5 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 27
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Lenses With Axis Orientation Within ±30 Degrees From the 90 Degree Axis (Ideal Location)
Description: Each lens was classified based on whether the absolute difference between the axis location and 90° was less than or equal to 30° (ie, lens axis located between the 60° and 120° axis inclusive). Inferential testing was not planned for this primary effectiveness endpoint.
Time Frame: Day 1, 10 minutes after lens insertion, each product
Population: Full Analysis Set
Measure: Number; unit: percentage of lenses
Units Other Than Participants: Eyes
Groups:
- AOHG Toric: Lotrafilcon B toric contact lenses with HYDRAGLYDE® worn in both eyes for approximately 30 minutes during either Period 1 or Period 2, as randomized
- AO Toric: Lotrafilcon B toric contact lenses worn in both eyes for approximately 30 minutes in either Period 1 or Period 2, as randomized
Arm/Group | AOHG Toric | AO Toric
Number analyzed (Participants) | 36 | 36
Number analyzed (Eyes) | 72 | 72
percentage of lenses | 94.4 | 95.8

ADVERSE EVENTS:
Time Frame: Dispense through study completion, approximately 2 hours
Description: An adverse event (AE) was defined as any untoward medical occurrence, unintended disease or injury, or untoward clinical signs in subjects, users, or other persons, whether or not related to the investigational medical device. AEs were obtained through solicited and spontaneous comments from subjects and through observations by the Investigator as outlined in the protocol. This analysis population includes all subjects/eyes exposed to any study lenses evaluated.
Groups:
- AOHG Toric: All subjects exposed to lotrafilcon B toric contact lenses with HYDRAGLYDE® in Period 1 or Period 2, as randomized
- AO Toric: All subjects exposed to lotrafilcon B toric contact lenses in Period 1 or Period 2, as randomized
Arm/Group | AOHG Toric | AO Toric
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/36
Other Adverse Events (participants affected / at risk) | 0/36 | 0/36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.

DOCUMENTS (2):
  • Study Protocol (2017-11-17): https://cdn.clinicaltrials.gov/large-docs/32/NCT03392532/Prot_000.pdf
  • Statistical Analysis Plan (2017-12-11): https://cdn.clinicaltrials.gov/large-docs/32/NCT03392532/SAP_001.pdf